CLINICAL TRIAL: NCT07140692
Title: VISTA OPHTHALMICS 1-STEP VITRECTOR POST MARKET LIMITED VITREOUS REMOVAL (LVR) CLINICAL ASSESSMENT
Brief Title: EFFECTIVENESS AND SAFETY ASSESSMENT OF THE VISTA VITRECTOMY PROBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Centers of Racine and Kenosha (Other)
Responsible Party: Principal Investigator, Inder Paul Singh, M.D., Ophthalmologist and President, The Eye Centers of Racine & Kenosha, The Eye Centers of Racine and Kenosha
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECRK-LVR-01
Record Dates: First submitted 2025-08-22; First posted 2025-08-25 (Actual); Last update posted 2025-08-25 (Actual); Status verified 2025-08

CONDITIONS: Vitreous Floaters; Vitreous Opacities
Keywords: Vitrectomy; Vista 1-Step Vitrector; Vitreous opacities or floaters
MeSH Terms: conditions — vitreous floaters | interventions — Vitrectomy

STUDY DESIGN:
Intervention Model Description: The Vista Ophthalmics 1-Step Vitrector is intended to perform anterior/posterior vitrectomy procedures and remove vitreous and dissected tissue in the eye. It consists of a single-use vitrector with air supply tubing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vista Ophthalmics vitrectomy (Experimental): In this single-arm, non-comparative study, patients presenting with vitreous opacities affecting daily activities of living will undergo vitrectomy using the single-use vitrector probe of Vista Ophthalmics for the removal of the vitreous opacities.
  Interventions: Device: Vitrectomy

INTERVENTIONS:
Device: Vitrectomy — In this single-arm, non-comparative study, patients presenting with vitreous opacities affecting daily activities of living will undergo vitrectomy using the single-use vitrector probe of Vista Ophthalmics for the removal of the vitreous opacities.

SUMMARY:
Vitreous opacities or floaters are a common ocular condition that can cause significant impairment in vision-related quality of life (QoL) in some patients. Vitrectomy involves the surgical removal of vitreous humour, the transparent jelly, from inside the eye that contains vitreous opacities and floaters. The present post-market clinical assessment study aims to assess the safety and effectiveness performance of the Vista 1-Step vitrectomy probe in adult pseudophakic patients with visually symptomatic opacities.

DETAILED DESCRIPTION:
Vitreous opacities or floaters are a common ocular condition that seems ubiquitous in a retina practice. Although symptoms are minimal in most patients, they can cause significant impairment in vision-related quality of life (QoL) in some patients.

Vitrectomy is a surgical procedure to remove the vitreous humour, the transparent jelly, from inside the eye. Vitrectomy Surgery can be of two types: Full and Limited. Full Vitrectomy is the commonly used and standard technique for repairing retinal detachments, removing membranes or haemorrhages, and involves vitreous detachment from the retina and its removal, both centrally and peripherally. Limited Vitrectomy is a new technique which focuses on the removal of only the central part of the vitreous or Core with the Vitreous Opacities or "Floaters" in it, and without intentionally detaching it from the retina.

The Vista Ophthalmics vitrectomy probe is a single-use vitrector intended to perform anterior/posterior vitrectomy procedures and to remove vitreous and dissect tissue in the eye. The Vista Ophthalmic's probe is designed as a stand-alone handpiece for use with ophthalmic systems.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant with age ≥ 18 years at the time of screening.
2. Subjects with Posterior chamber Intraocular lens (PCIOL) in one or both the eyes (both eyes will be independently assessed).
3. Subjects must be able to understand and voluntarily provide written informed consent before screening, following an explanation of the nature and purpose of this study.
4. Subjects must be willing and able to comply with all treatment and follow-up study procedures.
5. Complaints of decreased vision/decreased quality of vision due to vitreous floaters which is having an impact on Activities of daily living (ADLs).
6. Documentation of vitreous opacities on Slit lamp exam/Dilated Fundus Exam (SLE/DFE).
7. Documentation of decreased DLI on iTrace.

Exclusion Criteria:

1. Subjects with history of retinal tear/detachment, macular edema, Epi-retinal membrane (ERM), vitreomacular traction syndrome (VMT), Age-related macular degeneration (AMD), Proliferative Diabetic Retinopathy (PDR), or other significant retinal disorders in procedural eye.
2. Subjects with History of trauma to operative eye.
3. Subjects with bleeding disorders or anticoagulation.
4. Subjects with history of ocular herpetic infections.
5. Female subjects of child bearing potential with positive urine pregnancy test.
6. Subjects who have participated in any drug or device clinical investigation within 30 days prior to entry into or during this study.
7. Any medical condition that would be contraindicated for cataract surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Degree of change in iTrace Dysfunctional Lens Index (DLI) from baseline to post-operative visit Day 30 | Day 30 (+/- 7 days)
  iTrace Dysfunctional Lens Index (DLI) score
Degree of change in Kim Floater Survey from baseline to post-operative visit Day 30 | Day 30 (+/-7 days)
  Assessment using Kim Floater Questionnaire
Degree of change in surgeon assessed vitreous opacities from baseline to post-operative visit Day 30 | Day 30 (+/-7 days)
  Dilated Fundus/Peripheral Exam

SECONDARY OUTCOMES:
Incidence of post-operative adverse events | Day 30 (+/- 7 days)
  Ophthalmic examination

CONTACTS AND LOCATIONS:
Locations (1):
- The Eye Centers of Racine & Kenosha, Kenosha, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No